CLINICAL TRIAL: NCT03757559
Title: A Single-dose, Nested-randomized, Double-blind, Double-dummy, Placebo- and Active-controlled Crossover Trial to Evaluate the Abuse Potential of 3 Doses of GRT6005 in Adult Non-dependent Recreational Opioid Users
Brief Title: A Trial to Evaluate the Abuse Potential of 3 Doses of GRT6005 in Adult Non-dependent Recreational Opioid Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP6005/10
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Abuse, Drug
Keywords: Cebranopadol; Hydromorphone; Drug liking
MeSH Terms: conditions — Substance-Related Disorders | interventions — Hydromorphone

STUDY DESIGN:
Intervention Model Description: Nested-randomized, single site, double-blind, double-dummy, placebo- and active-controlled, crossover design with administration of a single oral dose. Based on the assigned treatment sequence, each participant was randomly allocated to receive a single oral dose of the investigational medicinal product (IMP) in each of 7 periods. One administration of placebo (Treatment G) always followed cebranopadol 800 micrograms (Treatment C). Each IMP administration was given under fasted conditions and was separated by a washout period of at least 14 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cebranopadol 200 micrograms (Treatment A) (Experimental): Cebranopadol 200 micrograms (low dose): Participants took 2 tablets (cebranopadol 100 micrograms) as a single dose.
  In addition, participants took 4 placebo capsules matching hydromorphone capsules as a single dose.
  Interventions: Drug: Cebranopadol 100 micrograms; Drug: Placebo matching hydromorphone
- Cebranopadol 400 micrograms (Treatment B) (Experimental): Cebranopadol 400 micrograms (medium dose): Participants took 2 tablets (cebranopadol 400 micrograms plus matching placebo) as a single dose.
  In addition, participants took 4 placebo capsules matching hydromorphone capsules as a single dose.
  Interventions: Drug: Cebranopadol 400 micrograms; Drug: Placebo matching hydromorphone
- Cebranopadol 800 micrograms (Treatment C) (Experimental): Cebranopadol 800 micrograms (high dose): Participants took 2 tablets containing cebranopadol 400 micrograms as a single dose.
  In addition, participants took 4 placebo capsules matching hydromorphone capsules as a single dose.
  Interventions: Drug: Cebranopadol 400 micrograms; Drug: Placebo matching hydromorphone
- Hydromorphone IR 8 milligrams (Treatment D) (Active Comparator): Hydromorphone immediate-release (IR) 8 milligrams: Participants took 4 capsules (2 capsules of hydromorphone hydrochloride 4 mg plus 2 placebo capsules) as a single dose.
  In addition, participants took 2 placebo tablets matching cebranopadol tablets as a single dose.
  Interventions: Drug: Hydromorphone hydrochloride 4 milligrams; Drug: Placebo matching cebranopadol
- Hydromorphone IR 16 milligrams (Treatment E) (Active Comparator): Hydromorphone immediate-release (IR) 16 milligrams: Participants took 4 capsules of hydromorphone hydrochloride 4 mg as a single dose.
  In addition, participants took 2 placebo tablets matching cebranopadol tablets as a single dose.
  Interventions: Drug: Hydromorphone hydrochloride 4 milligrams; Drug: Placebo matching cebranopadol
- Placebo (Treatment F) (Placebo Comparator): Placebo: Participants took 4 placebo capsules matching hydromorphone capsules as a single dose.
  In addition, participants took 2 placebo tablets matching cebranopadol tablets as a single dose.
  Interventions: Drug: Placebo matching hydromorphone; Drug: Placebo matching cebranopadol
- Placebo (Treatment G) (Placebo Comparator): Placebo (following Treatment C): Participants took 2 placebo tablets matching cebranopadol tablets as a single dose.
  In addition, participants took 4 placebo capsules matching hydromorphone capsules as a single dose.
  Interventions: Drug: Placebo matching hydromorphone; Drug: Placebo matching cebranopadol

INTERVENTIONS:
Drug: Cebranopadol 100 micrograms — Tablets were taken under fasted conditions with non-carbonated water.
  Arms: Cebranopadol 200 micrograms (Treatment A)
Drug: Cebranopadol 400 micrograms — Tablets were taken under fasted conditions with non-carbonated water.
  Arms: Cebranopadol 400 micrograms (Treatment B); Cebranopadol 800 micrograms (Treatment C)
Drug: Hydromorphone hydrochloride 4 milligrams — Over-encapsulated immediate-release tablets were taken under fasted conditions with non-carbonated water.
  Other Names: Dilaudid (Trade Mark) 4 mg
  Arms: Hydromorphone IR 16 milligrams (Treatment E); Hydromorphone IR 8 milligrams (Treatment D)
Drug: Placebo matching hydromorphone — Placebo matching over-encapsulated hydromorphone tablets were taken under fasted conditions with non-carbonated water.
  Arms: Cebranopadol 200 micrograms (Treatment A); Cebranopadol 400 micrograms (Treatment B); Cebranopadol 800 micrograms (Treatment C); Placebo (Treatment F); Placebo (Treatment G)
Drug: Placebo matching cebranopadol — Placebo matching cebranopadol tablets were taken under fasted conditions with non-carbonated water.
  Arms: Hydromorphone IR 16 milligrams (Treatment E); Hydromorphone IR 8 milligrams (Treatment D); Placebo (Treatment F); Placebo (Treatment G)

SUMMARY:
The primary objective of this study was to evaluate the abuse potential of single doses of cebranopadol (GRT6005) relative to hydromorphone (immediate-release formulation [IR] and placebo in 48 non-dependent recreational opioid users.

Secondary objectives were to evaluate the abuse potential of hydromorphone IR compared to placebo (trial validation), to evaluate the safety and tolerability of single doses of cebranopadol (200, 400, and 800 micrograms), and to evaluate pharmacokinetics (PK) of cebranopadol and optionally some of its metabolites.

DETAILED DESCRIPTION:
The study comprised an Enrollment Visit, a Qualification Phase, a Treatment Phase with 7 double-blind treatment periods for each participant, and a Final Examination.

In the Qualification Phase, all participants completed a naloxone challenge test to confirm that they were not opioid-dependent. The Objective Opioid Withdrawal Scale was used to record the signs or symptoms of withdrawal observed during the naloxone challenge test. Following the naloxone challenge test, participants received a single oral dose of hydromorphone immediate-release (IR) 12 milligrams (mg) and placebo in a double-blinded, randomized crossover manner to ensure that they could discriminate between an active drug and placebo and could tolerate hydromorphone IR 12 mg. After a washout phase of at least 3 days, participants could continue with the Treatment Phase.

In the Treatment Phase, each participant received single oral doses of the 7 different investigational medicinal products (IMPs) (Treatment A to Treatment G) in 7 sequential treatment periods. The treatment sequences per participant were randomly assigned, except for one administration of placebo (Treatment G) which always followed the highest dose of cebranopadol (Treatment C). Each IMP administration was given under fasted conditions and was separated by a washout period of at least 14 days.

Participants were confined to the study site from Day -1 until 48 hours after the first IMP administration in the Qualification Phase and from Day -1 until 56 hours after the IMP administration in the treatment periods. Pharmacodynamic assessments and blood sampling for pharmacokinetics were performed from pre-dose until 56 hours post-dose in each treatment period.

The Final Examination was conducted 5 days to 10 days after the discharge from the last treatment period or upon early discontinuation from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed.
2. Male and female, aged 18 years to 55 years, inclusive.
3. History of recreational opioid use (defined as non-therapeutic use at least 10 times in the participant's lifetime and at least once in the last 12 weeks prior to the Enrollment Visit).
4. Body mass index between 19 kilograms per square meter and 32 kilograms per square meter inclusive, with a body weight of not less than 50 kilograms at enrollment.
5. Participants must be in good health as determined by medical history, physical examination, 12-lead electrocardiogram (ECG), and vital signs (pulse rate, systolic blood pressure and diastolic blood pressure, respiratory rate, and oxygen saturation using pulse oximetry) at enrollment.
6. Adequate contraception is being used or women of non-childbearing potential may be enrolled if surgically sterile (i.e., after hysterectomy) or post-menopausal for at least 2 years (based on participant's report).

   * For women of childbearing potential: A medically acceptable and highly effective method of birth control is defined as any form of contraception with a low failure rate defined as less than 1 percent per year. For example:

     * Hormonal contraceptives for at least 8 weeks prior to the Enrollment Visit and at least until 4 weeks after the Final Examination.
     * An intra-uterine device. Additional barrier contraception should be used by the partner for the duration of the study, defined as from the time of the Enrollment Visit until 4 weeks after the Final Examination. A single barrier method alone is not acceptable.
   * For men: Participants must be willing to use medically acceptable and highly effective methods of birth control. Participants must be willing to use barrier contraception (condom) during sexual intercourse with females from the first administration of investigational medicinal product (IMP) until 4 weeks after the Final Examination. Participants must be willing to take care that their female sexual partner uses at least 1 additional method of contraception with a low failure rate defined as less than 1 percent per year (e.g., hormonal contraceptives, diaphragm) during this time frame. A single barrier method alone is not acceptable.

Exclusion Criteria (at Enrollment):

1. Current substance dependence (except nicotine and caffeine dependence) as defined by the Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV).
2. Unwillingness or inability to abstain from recreational drug use for the duration of the study.
3. Positive or missing alcohol breath test at enrollment.
4. Participants attempting to discontinue their recreational drug use or who had been in a drug rehabilitation program in the 12 months prior to enrollment.
5. Current consumption of more than 20 cigarettes per day or inability to abstain from smoking (or use of any nicotine-containing substance) for at least 26 hours.
6. Participation in another clinical study within 30 days prior to enrollment that resulted in the administration of at least 1 dose of IMP.
7. Diseases or conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
8. Prolongation of corrected QT interval (Fridericia) (QTcF) (after repeated assessment) at enrollment, i.e., above 450 milliseconds, or presence of additional risk factors for torsade de pointes (e.g., heart failure, hypokalemia), or use of concomitant medications that prolong QT interval.
9. History of orthostatic hypotension or other cardiovascular diseases.
10. Any clinically significant disease that in the investigator's opinion may affect efficacy or safety assessments or may compromise the participant's safety during study participation, e.g., significant pulmonary, gastrointestinal, cardiac, endocrine, metabolic, neurological, or psychiatric disorders.
11. Definite or suspected history of drug allergy or hypersensitivity to opioids or naloxone.
12. Use of forbidden medication within 2 weeks prior to enrollment into this study.
13. Any contraindication for naloxone or hydromorphone immediate-release (IR) administration.
14. Not able to abstain from consumption of:

    * Beverages or food containing caffeine (tea, coffee, cola, chocolate, etc.) or alcohol from 2 days prior to each Day 1 until discharge from the ward.
    * Beverages or food containing quinine (e.g., bitter lemon, tonic water) from 1 week before Day 1 of the Qualification Phase until the Final Examination.
    * Grapefruit juice (sweet or sour) or Seville oranges from 1 week before Day 1 of the Qualification Phase until the Final Examination.
15. Pregnant or breastfeeding women, or missing pregnancy test.
16. Blood loss of 500 milliliters or more within 4 weeks before enrollment in this study, including blood donation. Planned blood donations during the study and up to 12 weeks after the Final Examination.
17. History of seizure disorder and/or epilepsy or any condition associated with a significant risk for seizure disorder or epilepsy at the Enrollment Visit at the discretion of the investigator.
18. Known or suspected of not being able to comply with the study protocol.
19. Not able to communicate meaningfully with the investigator or study site staff.
20. Employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator.

Exclusion criteria (for Day 1) (Qualification Phase):

1. Positive naloxone challenge on Day -1 of the Qualification Phase.
2. Use of forbidden medication since the Enrollment Visit
3. Positive or missing urine pregnancy test.
4. Positive or missing alcohol breath test.
5. Positive or missing urine drug of abuse screen result, except for cannabinoids (tetrahydrocannabinol [THC]; due to slow release from adipose), which must be negative, stable, or decreasing. If THC is not negative, stable, or decreasing, inclusion will be at the discretion of the investigator, in consultation with the sponsor.
6. Positive or missing viral serology, i.e., human immunodeficiency virus Type 1 and Type 2 antibodies and antigen, hepatitis B surface antigens, antibodies to hepatitis B core antigen and immunoglobulin M antibody to hepatitis B core antigen, and hepatitis C virus antibodies, based on sample taken at the Enrollment Visit.
7. Any abnormal laboratory values or any clinically relevant out-of-range values for safety laboratory parameters (clinical chemistry, clotting, hematology, and urinalysis) based on sample taken at the Enrollment Visit, as judged by the investigator.
8. Blood donation or acute loss of blood (more than 100 milliliters) since the enrollment excluding blood samples required by the protocol.
9. Any relevant deterioration in the health of the participant that could alter the benefit/risk assessment for the participant, including adverse events, laboratory parameters, vital signs, or other safety parameters (e.g., ECGs).
10. Failure to comply with study requirements, e.g., intake of forbidden medications, consumption of alcohol, etc., considered by the investigator to affect participant safety or interfere with the integrity of the study.
11. Uncooperative participants or participants who refused to continue in the study.
12. Withdrawal of informed consent.
13. Any contraindication for naloxone or hydromorphone IR administration.

Discontinuation criteria for Day 1 (Treatment Phase):

1. Failure to successfully fulfill any of the following criteria based on the qualification period prior to the first treatment period (Treatment Period 1, Day -1):

   * Peak scores (Emax) in response to hydromorphone greater than that of placebo on (at this moment) Drug Liking VAS (difference of at least 15 points).
   * Acceptable responses to placebo and hydromorphone on visual analog scale (VAS) for (at this moment) Drug Liking, High, Good Effects, Overall Drug Liking, Take Drug Again, and Feeling Sick, as judged by the investigator or designee and sponsor.
   * The ability to tolerate hydromorphone, as judged by the investigator based on available safety data (e.g., respiratory rate greater than or equal to 8 breaths per minute and no vomiting).
   * General behavior suggestive that they could successfully complete the study, as judged by the investigator.
2. Positive or missing urine pregnancy test.
3. Positive or missing alcohol breath test.
4. If a participant tests positive for other drugs of abuse, the urine drug screen can be repeated and/or the participant rescheduled at the discretion of the investigator or designee, in consultation with the sponsor.
5. Blood donation or acute loss of blood (more than 100 milliliters) since the Enrollment Visit excluding blood samples required by the protocol.
6. Any relevant deterioration in the health of the participant that could alter the benefit/risk assessment for the participant, including adverse events, laboratory parameters, vital signs, or other safety parameters (e.g., ECG).
7. Failure to comply with study requirements, e.g., intake of forbidden medications, consumption of alcohol, etc., considered by the investigator to affect participant safety or interfere with the integrity of the study.
8. Uncooperative participants or participants who refused to continue in the study.
9. Withdrawal of informed consent.
10. Not able to use adequate contraception as defined in Inclusion Criterion 6.
11. Not able to abstain from consumption of:

    * Beverages or food containing quinine (e.g., bitter lemon, tonic water).
    * Grapefruit juice (sweet or sour) or Seville oranges.
    * Beverages or food containing caffeine (tea, coffee, cola, chocolate, etc.) or alcohol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 226 (Actual)
Dates: Start 2013-04-15 (Actual); Primary Completion 2014-03-08 (Actual); Study Completion 2014-03-08 (Actual)

PRIMARY OUTCOMES:
Drug Liking (at this moment) | At 16 distinct time points between 30 minutes and 56 hours after drug intake
  Visual analog scale (VAS) rating; Question text: At this moment, my liking for this drug is ...; Bipolar response anchors: 0 (Strong disliking), 50 (Neither like nor dislike), 100 (strong liking).

SECONDARY OUTCOMES:
Any Drug Effects | At 16 distinct time points between 30 minutes and 56 hours after drug intake
  Visual analog scale (VAS) rating; Question text: I can feel any drug effect. Unipolar response anchors: 0 (Definitely not) to 100 (Definitely so).
Good Drug Effects | At 16 distinct time points between 30 minutes and 56 hours after drug intake
  Visual analog scale (VAS) rating; Question text: I can feel good drug effects; Unipolar response anchors: 0 (Definitely not) to 100 (Definitely so).
Bad Drug Effects | At 16 distinct time points between 30 minutes and 56 hours after drug intake
  Visual analog scale (VAS) rating; Question text: I can feel bad drug effects; Unipolar response anchors: 0 (Definitely not) to 100 (Definitely so).
High | Pre-dose and at 16 distinct time points between 30 minutes and 56 hours after drug intake
  Visual analog scale (VAS) rating; Question text: I am feeling high; Unipolar response anchors: 0 (Definitely not) to 100 (Definitely so).
Take Drug Again | At 12, 24, and 56 hours aft drug intake
  Visual analog scale (VAS) rating; Question text: I would take this drug again; Unipolar response anchors: 0 (Definitely not) to 100 (Definitely so).
Feeling Sick | Pre-dose and at 16 distinct time points between 30 minutes and 56 hours after drug intake
  Visual analog scale (VAS) rating: Question text: I am feeling sick; Unipolar response anchors: 0 (Definitely not) to 100 (Definitely so).
Alertness/Drowsiness | Pre-dose and at 16 distinct time points between 30 minutes and 56 hours after drug intake
  Visual analog scale (VAS) rating; Question text: My mental state is...; Bipolar response anchors: 0 (Very drowsy), 50 (Neither drowsy nor alert), 100 (Very alert).
Floating | Pre-dose and at 16 distinct time points between 30 minutes and 56 hours after drug intake
  Visual analog scale (VAS) rating; Question text: I feel as if I am floating; Unipolar response anchors: 0 (Not at all) to 100 (Very much).
Detached | Pre-dose and at 16 distinct time points between 30 minutes and 56 hours after drug intake
  Visual analog scale (VAS) rating; Question text: I feel detached from my body; Unipolar response anchors: 0 (Not at all) to 100 (Very much).
Overall Drug Liking | At 12, 24, and 56 hours aft drug intake
  Visual analog scale (VAS) rating; Question text: Overall, my liking for this drug is ...; Bipolar response anchors: 0 (Strong disliking), 50 (Neither like nor dislike), 100 (Strong liking)
Drug Similarity | At 12, 24, and 56 hours aft drug intake
  Visual analog scale (VAS) rating; Questions 1-15: How similar is the drug you most recently received to...? with 15 drugs to be assessed and response anchors 0 (Not at all similar) to 100 (Very similar); Question 16: How familiar was the effect of the drug you most recently received? for an overall familiarity assessment with response anchors 0 (Very unfamiliar) to 100 (Very familiar).
Morphine-Benzedrine Group (MBG) scale | Pre-dose and at 16 distinct time points between 30 minutes and 56 hours after drug intake
  The Addiction Research Center Inventory (ARCI) scale to assess euphoria (MBG scale) was presented to the participant on a computer screen as multiple choices. Participants were asked to select their responses by pointing to one of them with the mouse; the two responses are "False" or "True".
Benzedrine Group (BG) scale | Pre-dose and at 16 distinct time points between 30 minutes and 56 hours after drug intake
  The Addiction Research Center Inventory (ARCI) scale to assess stimulant-like effects: amphetamine, A-scale and Benzedrine Group (BG scale) was presented to the participant on a computer screen as multiple choices. Participants were asked to select their responses by pointing to one of them with the mouse; the two responses are "False" or "True".
Pentobarbital-Chlorpromazine-Alcohol Group (PCAG) scale | Pre-dose and at 16 distinct time points between 30 minutes and 56 hours after drug intake
  The Addiction Research Center Inventory (ARCI) scale to assess sedation was presented to the participant on a computer screen as multiple choices. Participants were asked to select their responses by pointing to one of them with the mouse; the two responses are "False" or "True".
Pupillometry | Pre-dose and at 9 distinct time points between 1 and 56 hours after drug intake
  Pupil diameter was measured under mesopic lighting conditions. Data from a series of frames were used in the calculation, and the weighted average and standard deviation of the pupil size was calculated.
Divided Attention Test | Pre-dose and at 8 distinct time points between 1 and 56 hours after drug intake
  Manual-tracking test with a simultaneous visual target detection component. Participant is provided with joystick and presented with the image of an airplane and a randomly curving road; participant has to position the airplane over the center of the road while being distracted repeatedly by visual targets they have to respond to. Time over the road (percentage), response latency of correct responses (milliseconds) and target hits (percentage) are recorded.

OTHER OUTCOMES:
Area under the concentration-time curve up to the sampling time t (AUC0-t) | From pre-dose until 56 hours post-dose in each treatment period (13 samples in total)
  Plasma concentrations were determined using validated liquid chromatography-tandem mass spectrometry bioanalytical assays. Blood samples for pharmacokinetic analyses of cebranopadol and 3 of its metabolites were collected from pre-dose until 56 hours post-dose in each treatment period. The AUC0-t was calculated based on plasma concentration-time data (using the actual blood sampling times).
Time to attain maximum concentration (tmax) | From pre-dose until 56 hours post-dose in each treatment period (13 samples in total)
  Plasma concentrations were determined using validated liquid chromatography-tandem mass spectrometry bioanalytical assays. Blood samples for pharmacokinetic analyses of cebranopadol and 3 of its metabolites were collected from pre-dose until 56 hours post-dose in each treatment period. Tmax was calculated based on plasma concentration-time data (using the actual blood sampling times).
Maximum observed plasma concentration (Cmax) | From pre-dose until 56 hours post-dose in each treatment period (13 samples in total)
  Plasma concentrations were determined using validated liquid chromatography-tandem mass spectrometry bioanalytical assays. Blood samples for pharmacokinetic analyses of cebranopadol and 3 of its metabolites were collected from pre-dose until 56 hours post-dose in each treatment period. Cmax was calculated based on plasma concentration-time data (using actual blood sampling times).

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- INC Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No